CLINICAL TRIAL: NCT02524093
Title: The Efficacy of Positive Mental Training in Patients With Multiple Sclerosis Experiencing Psychological Distress: A Pilot Randomised Controlled Trial
Brief Title: The Impact of Positive Mental Training in Multiple Sclerosis
Acronym: PosMTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Principal Investigator, Katy Murray, Consultant Neuologist, University of Edinburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PosMT1.0
Record Dates: First submitted 2015-08-10; First posted 2015-08-14 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Multiple Sclerosis; Psychological Distress
MeSH Terms: conditions — Multiple Sclerosis | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in this arm will be given the Positive Mental Training programme. This consists of twelve eighteen minute audio tracks. Each is listened to in turn every day, once a day for a week (or at least 5 days in a week). This means that to use the treatment properly the participant needs to spend 18 minutes a day for 12 weeks listening to it. Each track guides the listener through different instructions which aim to build skills and bring about positive change. The programme begins with simple relaxation, going on to support the creation of pictures in your head of safe places and a more positive future.
  Interventions: Behavioral: Positive Mental Training
- Control (Placebo Comparator): Will receive treatment as usual for 12 weeks, when will be asked to complete rating scales again. They will then be given the Positive Mental Training programme.
  Interventions: Other: treatment as usual

INTERVENTIONS:
Behavioral: Positive Mental Training — Positive Mental Training consists of twelve eighteen minute audio tracks. Each is listened to in turn every day, once a day for a week (or at least 5 days in a week). This means that to use the treatment properly you need to spend 18 minutes a day for 12 weeks listening to it. Each track guides the listener through different instructions which aim to build skills and bring about positive change. The programme begins with simple relaxation, going on to support the creation of pictures in your head of safe places and a more positive future.
  Arms: Intervention
Other: treatment as usual
  Arms: Control

SUMMARY:
Depression and anxiety are common in MS and often go untreated. Even symptoms which do not meet the threshold for a psychiatric diagnosis can have a significant impact on quality of life. Positive Mental Training (PosMT) is a 12 week programme which aims to help people overcome the negative thinking and feelings that come with worry and low mood and become more positive, confident and resilient. To find out if Positive Mental Training is helpful in MS the investigators are running a randomised controlled trial. The initial study is a pilot tiral, the primary function being examination of the feasibility and acceptability of this treatment in MS. Though sample size is small and consequently it may not be powered to detect a significant change in symptoms in association with the treatment, this will also be examined.

DETAILED DESCRIPTION:
Psychiatric disturbance is common in multiple sclerosis (MS), with anxiety and depression the most frequent diagnoses. The lifetime rate of major depression is up to 50%. However, even symptoms of mood and anxiety which are not severe enough to warrant a diagnosis of a psychiatric disorder can still have a big impact people's lives. The investigators want to find ways to make people with MS feel better and cope better in their day to day life, and to be stronger inside themselves so that they don't become worried or stressed so much in the future. Positive Mental Training (PosMT) is a 12 week programme which aims to help people overcome the negative thinking and feelings that come with worry and low mood and become more positive, confident and resilient. To find out if Positive Mental Training is helpful in MS the investigators are running randomised controlled trial. Patients with MS who score higher than 4 on either the Hospital Anxiety (HADS-A) or Depression Scale (HADS-D) will be admitted to the trial. They will be randomly allocated to either an intervention or control group. The intervention group will be given the treatment immediately, the other 12 weeks later. In addition to the HADS, patients will be asked to complete two further questionnaires asking about how low mood and anxiety affecting them, both when they enter the trial and 12 weeks later. These are the Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS) and EuroQol health related quality of life - 5 dimensions - 5 levels (EuroQol-5D-5L). The primary function of this pilot trial is to ascertain suitability and acceptability of this treatment for people with MS, and to guide planning of a subsequent full trial. Feedback will therefore be obtained from participants in the treatment group of their experience of using the intervention. Though the sample size of this pilot trial is small, by comparing the change in scores on rating scales in patients given the treatment to those who have not been given it yet (the control group), it may be feasible to ascertain if PosMT is a useful treatment in MS.

ELIGIBILITY:
Inclusion Criteria:

* Have confirmed diagnosis of Multiple Sclerosis

Exclusion Criteria:

* Lack capacity to provide informed consent
* Judged by the treating clinician to have cognitive deficits of such severity to preclude engagement with the treatment
* Felt by the treating clinician to be unsuitable to participate on other clinical grounds (e.g. significant receptive aphasia) will be excluded.
* Do not speak English (they would be unable to independently make use of the intervention)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Change from baseline after 12 weeks
Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS) | Change from baseline after 12 weeks

SECONDARY OUTCOMES:
Assessment of health-related quality of life - EuroQol health related quality of life - 5 dimensions - 5 levels (EuroQol-5D-5L) | Change from baseline after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katy Murray, MD, Principal Investigator — NHS Lothian
Locations (1):
- Anne Rowling Clinic, Edinburgh, Scotland, United Kingdom